CLINICAL TRIAL: NCT07356401
Title: Association Between Cranial Morphological Changes, Parental Expectations, and Satisfaction Following Cranial Remolding Orthosis Treatment in Infants
Brief Title: Associations of Cranial Outcomes and Parental Expectations and Satisfaction
Status: Recruiting | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Güllü Aydın Yağcıoğlu, Asst. Prof, Gulhane School of Medicine
Other Study IDs: cranial orthosis
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-11

CONDITIONS: Plagiocephaly; Cranial Defect; Orthosis; Expectancy; Satisfaction
MeSH Terms: conditions — Plagiocephaly; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- infant with cranial deformity: Infants presenting with cranial deformities characterized by abnormal cranial shape or asymmetry during early infancy, including deformities affecting cranial symmetry, cranial proportions, and head contour. Participants are infants within the period of rapid cranial growth, for whom cranial remolding orthosis treatment is clinically indicated. The cohort includes infants of both sexes, with varying degrees of cranial deformity severity, and without neurological or syndromic conditions that could affect cranial growth. All infants are otherwise medically stable and suitable for conservative orthotic management.
  Interventions: Device: Cranial orthosis

INTERVENTIONS:
Device: Cranial orthosis — The intervention consisted of treatment with a custom-fabricated cranial remolding orthosis (CRO). Each orthosis was individually designed based on the infant's cranial shape using three-dimensional cranial scanning and computer-aided modeling. A mold was produced using CNC technology, and a thermoplastic material was formed over the mold to create the final orthosis. The fabricated CRO was delivered to the clinic within a few days and fitted to the infant.
  During the initial fitting, the orthosis was clinically inspected for proper fit and for any signs of skin redness, irritation, or pressure-related issues. Necessary adjustments were made, and parents were provided with detailed instructions regarding orthosis use and care. Infants were subsequently scheduled for regular clinical follow-up, and only custom-fabricated cranial remolding orthoses were included in the study.

SUMMARY:
This study aims to investigate the association between objective cranial morphological changes and parental expectations and satisfaction in infants undergoing treatment with a cranial remolding orthosis (CRO). Infants diagnosed with positional cranial deformities and prescribed CRO treatment will be included. Cranial morphological outcomes will be assessed using standardized cranial measurements obtained before and after the treatment period.

Parental treatment expectations will be evaluated prior to the initiation of CRO therapy using the Treatment Expectation Questionnaire (TR.TEX-Q), while parental satisfaction with the device and treatment process will be assessed at the end of treatment using the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST).

The primary objective of the study is to examine the relationships between changes in cranial morphology and parental expectations and satisfaction scores. Secondary objectives include exploring the association between baseline expectations and post-treatment satisfaction. The findings are expected to provide insight into how objective treatment outcomes align with family-reported perceptions in cranial remolding orthosis therapy.

ELIGIBILITY:
Inclusion Criteria:

* Infants diagnosed with positional cranial deformities (e.g., plagiocephaly, brachycephaly, or asymmetrical cranial shape)
* Infants who received cranial remolding orthosis treatment
* Use of a custom-made cranial remolding orthosis
* Availability of pre-treatment and post-treatment cranial measurements
* Parents or legal guardians who provided informed consent and were able to complete expectation and satisfaction questionnaires
* Infants who completed the planned cranial remolding orthosis treatment and follow-up period

Exclusion Criteria:

* Infants with neurological disorders, genetic syndromes, or congenital conditions affecting cranial growth
* Infants who underwent previous cranial surgery or other cranial interventions
* Infants who received non-custom-made or prefabricated cranial orthoses
* Incomplete clinical records or missing pre- or post-treatment cranial measurements
* Parents or caregivers unable to complete the questionnaires due to language or cognitive limitations
* Infants with a diagnosis of microcephaly or macrocéphaly.

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study includes infants aged 3-18 months with cranial deformities who have been recommended helmet therapy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in cranial morphological measurements following cranial remolding orthosis treatment | Periprocedural
  The primary outcome measure is the change in cranial morphology assessed by standardized anthropometric measurements obtained before and after cranial remolding orthosis (CRO) treatment. Cranial measurements include anterior-posterior and medio-lateral dimensions, right and left frontal measurements, and head circumference. Changes in these measurements are used to quantify objective cranial morphological improvement over the course of treatment.
Parental treatment expectations | baseline
  Parental expectations regarding cranial remolding orthosis treatment are assessed before initiation of treatment using the Treatment Expectation Questionnaire. This measure evaluates parents' expectations related to treatment outcomes, process, and perceived benefits prior to intervention.The Treatment Expectation Questionnaire is a generic, multidimensional patient-reported outcome measure consisting of 15 items assessing expectations across multiple domains of treatment. Each item is rated on a numerical scale from 0 (no expected change) to 10 (maximum expected change), yielding a total score range of 0 to 150, with higher scores indicating greater treatment expectations.

SECONDARY OUTCOMES:
Parental satisfaction | Periprocedural
  Parental satisfaction with cranial remolding orthosis treatment is assessed after completion of the treatment period using the Quebec User Evaluation of Satisfaction with Assistive Technology. This measure evaluates satisfaction with the cranial remolding orthosis in terms of device-related characteristics and overall satisfaction with the assistive technology.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Gülhane Faculty of Health Sciences, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee HS, Kim SJ, Kwon JY. Parents' Perspectives and Clinical Effectiveness of Cranial-Molding Orthoses in Infants With Plagiocephaly. Ann Rehabil Med. 2018 Oct;42(5):737-747. doi: 10.5535/arm.2018.42.5.737. Epub 2018 Oct 31. PMID 30404423
- [Result] McGarry A, Dixon MT, Greig RJ, Hamilton DR, Sexton S, Smart H. Head shape measurement standards and cranial orthoses in the treatment of infants with deformational plagiocephaly. Dev Med Child Neurol. 2008 Aug;50(8):568-76. doi: 10.1111/j.1469-8749.2008.03017.x. PMID 18754893